CLINICAL TRIAL: NCT07139600
Title: A Study of Multi-omics Changes in Aplastic Anemia Patients Receiving CD7-CAR-T Therapy
Brief Title: Multi-omics Profiling of Patients With Aplastic Anemia Before and After CD7-CAR-T Therapy
Status: Active, not recruiting | Type: Observational
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Kai Lin Xu，MD, Chief Hematologist of The Affiliated Hospital of Xuzhou Medical University, Xuzhou Medical University
Other Study IDs: XYFY2024-KL365-01
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Aplastic Anaemia; CAR-T; CD7 Positive
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: CD7 CAR-T cells infusion — Autologous T cells are collected by leukapheresis, activated, and transduced with a retroviral vector encoding a CD7-specific CAR. Following fludarabine/cyclophosphamide lymphodepletion, CD7-CAR-T cells (3 × 10^6/kg) are infused intravenously. This intervention is distinguished by its CD7 target, aiming to suppress aberrant T-cell-mediated marrow destruction and restore hematopoiesis in aplastic anemia.

SUMMARY:
Aplastic anemia (AA) is a life-threatening bone marrow failure disorder characterized by pancytopenia and hypocellular bone marrow, with immune-mediated destruction of hematopoietic stem and progenitor cells (HSPCs) playing a central role in its pathogenesis. Although immunosuppressive therapy (IST) and hematopoietic stem cell transplantation (HSCT) have improved survival, a significant proportion of patients remain refractory, relapse after treatment, or lack suitable donors for transplantation. Therefore, novel therapeutic strategies are urgently needed.

Chimeric antigen receptor T (CAR-T) cell therapy has demonstrated remarkable efficacy in hematologic malignancies. CD7 is an early surface marker of T-lineage cells and is dispensable for T cell development and function, making it a promising therapeutic target. This exploratory study aims to investigate the molecular and cellular mechanisms of CD7-CAR-T therapy in AA patients by analyzing multi-omics changes before and after treatment.

This is a prospective, single-center, single-arm, open-label study enrolling patients with relapsed or refractory severe aplastic anemia. Participants will receive autologous CD7-CAR-T cells following lymphodepletion. Multi-omics profiling, including genomics, transcriptomics, proteomics, and immunophenotyping, will be performed on patient samples before and after infusion. The primary objective is to explore dynamic molecular changes associated with treatment response and disease progression. Secondary objectives include safety evaluation and preliminary assessment of efficacy.

Findings from this study may provide mechanistic insights into CD7-CAR-T therapy in AA and inform the development of innovative immunotherapies for bone marrow failure syndromes.

DETAILED DESCRIPTION:
This is a single-center, single-arm, prospective clinical study evaluating the safety and efficacy of CD7-directed CAR-T cell therapy in adult patients with refractory or relapsed severe aplastic anemia (SAA). SAA is an acquired bone marrow failure disorder characterized by pancytopenia and hypocellular marrow without malignant infiltration. Standard immunosuppressive therapy (IST) has improved survival, but approximately 30% of patients fail initial treatment, and relapse or progression to myelodysplastic syndrome or acute myeloid leukemia remains a clinical challenge. Allogeneic hematopoietic stem cell transplantation (allo-HSCT) improves outcomes for younger patients but is limited by donor availability and graft-versus-host disease risks.

Eligible participants are adults (≥18 years) with ECOG performance status 0-1, life expectancy ≥3 months, and refractory or relapsed SAA after IST, or ineligible for, lacking access to, or refusing allo-HSCT. Key laboratory criteria include creatinine ≤2.5× upper limit of normal, total bilirubin ≤3× ULN, ALT and AST ≤3× ULN, and baseline oxygen saturation ≥90%. Patients must have suitable venous access for leukapheresis and comply with contraception requirements if of reproductive potential. Exclusion criteria include active infections, severe cardiovascular disease, recent malignancy (except certain adequately treated cancers), pregnancy or breastfeeding, HIV, HBV, HCV above specified thresholds, or hypersensitivity to CAR-T components.

The study consists of four stages: patient screening and enrollment; preconditioning including leukapheresis, CAR-T cell manufacture, and chemotherapy; CD7-CAR-T cell infusion with inpatient monitoring; and long-term follow-up. Patients receive a lymphodepletion regimen with fludarabine and cyclophosphamide prior to a single infusion of CD7-CAR-T cells at 3×10^6 cells/kg. Safety assessments, including monitoring for cytokine release syndrome and other adverse events, will be conducted closely during hospitalization. Efficacy assessments include complete blood counts, bone marrow evaluation, and multi-omics analysis of immune cell subsets and cytokine profiles at defined intervals.

Participants will be followed up for up to 3 years post-infusion, with intensive monitoring in the first 6 months and periodic assessments thereafter to evaluate disease status, CAR-T cell persistence, long-term safety, and quality of life. The primary endpoint is overall response rate (ORR), with secondary endpoints including progression-free survival (PFS), overall survival (OS), and safety outcomes. This study aims to provide the first evaluation of CD7-CAR-T therapy in refractory or relapsed SAA patients, potentially offering a novel therapeutic option for this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years at the time of informed consent, of Chinese nationality. ECOG performance status 0-1, with an expected survival time ≥3 months.

Diagnosis of severe aplastic anemia (SAA) and meeting at least one of the following:

Relapsed or refractory after standard therapy without achieving complete remission.

Ineligible for, without access to, or refusing allogeneic hematopoietic stem cell transplantation.

Laboratory values at screening meeting all of the following:

Serum creatinine ≤2.5 × upper limit of normal (ULN). Oxygen saturation ≥90% at baseline. Total bilirubin ≤3 × ULN. ALT and AST ≤3 × ULN. Adequate venous access for mononuclear cell collection and no contraindications to leukapheresis.

Female participants of childbearing potential must have a negative high-sensitivity serum pregnancy test (β-hCG) at screening and before the first dose of fludarabine/cyclophosphamide. Male and female participants of childbearing potential must agree to use effective contraception from informed consent through at least 36 months after CD7-CAR-T infusion.

After review by the investigator team, the overall benefit of trial participation is judged to outweigh potential risks.

Ability to understand and sign informed consent, and willingness to comply with study procedures and restrictions.

Exclusion Criteria:

History of or treatment for other malignancies within 5 years prior to screening, except adequately treated cervical carcinoma in situ, basal or squamous cell skin cancer, curatively treated localized prostate cancer, or ductal carcinoma in situ.

Severe systemic diseases, including:

NYHA class III or IV congestive heart failure. Stroke, myocardial infarction, or hemodynamically unstable arrhythmia within 6 months prior to consent.

Left ventricular ejection fraction (LVEF) <50% by echocardiography. Severe or uncontrolled concomitant illness within 14 days prior to consent, including active infection.

Pregnant or breastfeeding women. Positive serology for HIV. Positive for hepatitis B surface antigen or detectable HBV DNA. Positive for hepatitis C antibody with detectable HCV RNA. Positive syphilis serology (TP-Ab and RPR). Positive CMV DNA.

History of life-threatening hypersensitivity to CD7-CAR-T cells or any excipients (including DMSO), or known hypersensitivity to biologics such as antibodies or cytokines.

Contraindications to fludarabine or cyclophosphamide therapy. History of alcohol dependence, substance abuse, or psychiatric disorders that may interfere with study compliance.

Any other condition that, in the opinion of the investigator, makes the participant unsuitable for the study.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) with refractory or relapsed severe aplastic anemia (SAA) after standard immunosuppressive therapy, or ineligible for/allogeneic hematopoietic stem cell transplantation. Participants must have ECOG 0-1, life expectancy ≥3 months, suitable venous access for leukapheresis, and meet basic lab criteria. Key exclusions include active infections, severe cardiovascular disease, recent malignancy, pregnancy/breastfeeding, or known HIV, HBV, or HCV infection.
Sampling Method: Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 36 months post-infusion.
  The proportion of patients achieving Complete Response (CR) or Partial Response (PR)
Progression-Free Survival (PFS) | Up to 36 months post-infusion.
  Time from CAR-T cell infusion to disease progression, relapse, or death from any cause, whichever occurs first.
Overall Survival (OS) | Up to 36 months post-infusion.
  Time from CAR-T cell infusion to death from any cause.
Event-Free Survival (EFS) | Up to 36 months post-infusion.
  Time from CAR-T cell infusion to the occurrence of any of the following events: failure to achieve response, disease progression or relapse, initiation of alternative therapy, or death from any cause.

SECONDARY OUTCOMES:
Safety and Tolerability | From infusion through study completion (up to 36 months).
  Incidence, severity, and type of treatment-emergent adverse events (TEAEs), including cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS). Graded according to CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Hai Cheng, Study Director — The Affiliated Hospital oh Xuzhou Medical University
Locations (1):
- Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No